CLINICAL TRIAL: NCT07205328
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase II Clinical Study to Evaluate the Efficacy and Safety of MT200605 in Patients With Acute Ischemic Stroke.
Brief Title: A Clinical Trial of MT200605 for the Treatment of Acute Ischemic Stroke
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shaanxi Micot Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MT200605-II-C01
Record Dates: First submitted 2025-09-25; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-07

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- MT200605 Low-dose group (Experimental): Standard medical treatment + MT200605 10mg, twice daily, intravenous infusion, for 14 consecutive days;
  Interventions: Drug: MT200605
- MT200605 Medium-dose group (Experimental): Standard medical treatment + MT200605 20mg, twice daily, intravenous infusion, for 14 consecutive days;
  Interventions: Drug: MT200605
- MT200605 High-dose group (Experimental): Standard medical treatment + MT200605 40mg, twice daily, intravenous infusion, for 14 consecutive days
  Interventions: Drug: MT200605
- Placebo Group (Placebo Comparator): Standard medical treatment + placebo, twice daily, intravenous infusion, for 14 consecutive days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MT200605 — MT200605 is an agonist of the receptor tyrosine kinase B (TrkB) and can enhances ATP synthesis in the mitochondria of the striatum and bolsters antioxidant and free radical-scavenging capabilities.
  Arms: MT200605 High-dose group
Drug: MT200605 — MT200605 is an agonist of the receptor tyrosine kinase B (TrkB) and can enhances ATP synthesis in the mitochondria of the striatum and bolsters antioxidant and free radical-scavenging capabilities.
  Arms: MT200605 Low-dose group
Drug: MT200605 — MT200605 is an agonist of the receptor tyrosine kinase B (TrkB) and can enhances ATP synthesis in the mitochondria of the striatum and bolsters antioxidant and free radical-scavenging capabilities.
  Arms: MT200605 Medium-dose group
Drug: Placebo — The placebo does not contain any active ingredients.
  Arms: Placebo Group

SUMMARY:
MT200605 is an agonist of the receptor tyrosine kinase B (TrkB). It exerts brain-derived neurotrophic factor (BDNF)-like effects, protecting the structure and function of neural tissues in the brain. Simultaneously, it enhances ATP synthesis in the mitochondria of the striatum and bolsters antioxidant and free radical-scavenging capabilities.

MT200605 is anticipated to confer pharmacological benefits including the reduction of neuronal apoptosis, antioxidant/free radical scavenging activity, anti-inflammatory effects, modulation of neuronal excitability, and amelioration of cerebral ischemic injury in patients with ischemic stroke.

This Phase II exploratory study will be conducted across 32 research centers in China. It plans to enroll 360 patients diagnosed with acute ischemic stroke within 24 hours of onset. Subjects will be randomized to receive either a high, medium, or low dose of MT200605 or a placebo, in addition to standard medical care. The primary efficacy endpoint is the proportion of subjects achieving a modified Rankin Scale (mRS) score of ≤1 at 3 months post-stroke. Secondary efficacy endpoints include the reduction in the National Institutes of Health Stroke Scale (NIHSS) score from baseline at day 14, among others.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 80 years old (inclusive), male or female ;
2. Diagnosed with ischemic stroke according to the "Chinese Guidelines for the Diagnosis and Treatment of Acute Ischemic Stroke 2023";
3. The time from the onset of the disease to the expected administration of the investigational drug will be within 24 hours., including patients who have not received reperfusion therapy or those have received intravenous thrombolysis treatment;
4. The NIHSS score at admission is between 6 and 25 (inclusive), and the sum of the scores for the 5th（upper limb movement） and the 6th（ lower limb movement） is ≥ 2 points;
5. The mRS score before this onset of stroke is 0 to 1, and there are no obvious clinical symptoms and signs that affect the NIHSS score;
6. Able to understand and cooperate with the process of this study, and voluntarily sign the informed consent.

Exclusion Criteria:

1. Imaging examinations show concurrent intracranial hemorrhagic disorders: such as hemorrhagic stroke, epidural hematoma, intracranial hematoma, ventricular hemorrhage, subarachnoid hemorrhage, etc. If there is minor bleeding, it could be determined based on the researcher's judgment whether the subject was suitable for inclusion;
2. After the onset of the disease, obvious consciousness disorders occurre, and the score of the NIHSS item for the 1a level of consciousness is >1 point;
3. Transient ischemic attack (TIA);
4. This acute ischemic stroke requires endovascular treatment (including intravenous thrombolysis, mechanical thrombectomy, angioplasty);
5. At the time of admission, already known severe active kidney disease, renal insufficiency; or serum creatinine > 1.5 × ULN;
6. Severe active liver diseases, such as acute hepatitis, chronic active hepatitis, liver cirrhosis, etc.; or ALT or AST > 2.0 × ULN;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin Scale（mRS） | 90 ± 5 days after the onset of stroke

CONTACTS AND LOCATIONS:
Locations (1):
- BeiJing Tiantan Hospital, Beijing, Beijing Municipality, China